CLINICAL TRIAL: NCT06473584
Title: Study of the Prevalence of Diabetes and Pre-diabetes in Réunion Island
Acronym: PREVADIABRUN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Collaborators: Agence Régionale de Santé de La Réunion (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023/CHU/42
Record Dates: First submitted 2024-06-19; First posted 2024-06-25 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Detection of glycaemic anomalies (Other)
  Interventions: Diagnostic Test: Diabetes detection

INTERVENTIONS:
Diagnostic Test: Diabetes detection — Fasting glycemia on blood sample

SUMMARY:
In view of the new priority given to diabetes in Réunion and the implementation of an ambitious plan to combat the disease at regional level, which includes the identification and management of pre-diabetes, the need for up-to-date data on the extent of these 2 diseases (diabetes and pre-diabetes) has become essential.

These two diseases have known risk factors: age, overweight, obesity, high waist circumference, family history, hypertension, eating habits and physical activity, all of which form part of a risk score for developing diabetes: the Findrisk recommended by the Haute Autorité de Santé for identifying people at risk of diabetes. Given the specific population characteristics of Réunion compared with Finland, where this score has been validated, it would seem important to be able to measure these risk indicators in the population as a function of carbohydrate status in order to check that the proposed thresholds are appropriate for the population of Réunion.

Finally, cardiovascular risk has been described as early as the pre-diabetes stage. Given the young age of onset of diabetes in Réunion and the high proportion of diagnoses of diabetes made following the occurrence of a cardiovascular complication, the study of the prognosis of carbohydrate status on the occurrence of complications using the social security information system will be offered on a voluntary basis to study subjects (via a probabilistic social security link).

ELIGIBILITY:
Inclusion Criteria:

* Have lived in Réunion island for at least one year
* Be aged between 18 and 75
* Affiliated to or benefiting from a social security scheme
* Free, informed and signed consent

Exclusion Criteria:

* No main residence on the island or fixed address for at least one year on the island
* Participation in experimental research
* Pregnant women
* Adults under guardianship or legal protection
* Not understanding French

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2025-04-02 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Estimating the prevalence of glycaemic abnormalities (diabetes and pre-diabetes) in Réunion | Day 1
  Measurement of fasting blood glucose and blood glucose 2 hours after ingesting 75g of glucose (HGPO test) according to Haute Autorite de Sante (HAS) recommendations used in France for diagnosing diabetes and pre-diabetes in people with unknown diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Catherine MARIMOUTOU, MD, PhD, Principal Investigator — CHU La Réunion
Locations (1):
- CHU La Réunion, Saint-Denis, Reunion